CLINICAL TRIAL: NCT06596148
Title: VA Quality Improvement Research and Training Initiative
Brief Title: Improving Shingrix Vaccination Among US Veterans Receiving Immunosuppression
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15-18358- SHINGRIX; I50HX003266 (NIH)
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Immunosuppresion
Keywords: Wait-list control randomized trial

STUDY DESIGN:
Intervention Model Description: The investigators will use a wait-list control design; clinicians from VA facilities will be randomized to receive access to the dashboard early vs. after a 6-9 month delay. The investigators will compare Shingrix vaccination rates in the two groups of facilities.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early dashboard access (Experimental): The early dashboard access arm will receive access to the Shingrix dashboard as soon as the study begins.
  Interventions: Other: Access to Shingrix dashboard
- Wait list control arm (Other): The wait list control arm will receive no intervention for 6-9 months; after this period, this arm will also receive access to the Shingrix dashboard.
  Interventions: Other: Access to Shingrix dashboard

INTERVENTIONS:
Other: Access to Shingrix dashboard — The investigators will build and grant access to a clinical dashboard that exists behind the VA firewall. The dashboard will identify Veterans from each VA facility who are receiving immunosuppressants (prescribed via the VA). The dashboard will also provide information about the number of Shingrix vaccines each patient has received (which have been documented within the VA electronic health record). VA clinicians will have access to view information about patients based on their VA electronic health record permissions.

SUMMARY:
The goal of this wait-list control trial is to learn if having access to a new dashboard displaying information about immunosuppressed Veterans missing vaccinations for Shingrix can improve Shingrix vaccination rates at VA facilities.

The main question[s] it aims to answer is: Will vaccination rates improve more rapidly for facilities with access to the dashboard compare to facilities without access? VA facility personnel will be granted access to the dashboard and outcomes (vaccination rates) will be measured using electronic health record data.

DETAILED DESCRIPTION:
Assignment of the intervention will occur at the facility level. Outcomes (vaccination) will be assessed for patients cared for at each facility.

ELIGIBILITY:
Inclusion Criteria:

* In order to be included in the study, clinicians need to work at a VHA facility and have access to the electronic health record.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with at least 1 Shingrix vaccine documented, by facility | From enrollment until end of follow up at 18 months.
  Percentage of patients with at least 1 Shingrix vaccinations documented, by facility

SECONDARY OUTCOMES:
Percentage of patients with at least 2 Shingrix vaccinations documented, by facility | From enrollment until end of follow up at 18 months.
  Percentage of patients with at least 2 Shingrix vaccinations documented, by facility

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Schmajuk, MD MS, Principal Investigator — San Francisco VA Medical Center
Locations (1):
- San Francisco VA, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
VA data is only available to VA investigators with specific permission under DUA.